CLINICAL TRIAL: NCT02700152
Title: Clinical Study to Evaluate the Safety and Efficacy of the UltraShape Device for Non-Invasive Abdominal Fat Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF18531
Record Dates: First submitted 2016-02-25; First posted 2016-03-07 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Excess Abdominal Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects (Experimental): Eligible subjects will receive 3 treatments, 2 weeks interval, with the UltraShape device according to the study protocol and user manual.
  The subject will return for 3 follow up visits: four weeks (4wk FU), eight weeks (8wk FU) and 12 weeks (12wk FU) after the last treatment, for total expected study duration of 16 weeks
  Interventions: Device: UltraShape

INTERVENTIONS:
Device: UltraShape — Tissue selectivity is achieved by a proprietary knowledge of ultrasound parameters ensuring specific destruction of the fat cells only within the target area. All other types of tissue, such as blood vessels, muscles and peripheral nerves remain intact. There are no thermal effects. Fat cell destruction is achieved by ultrasound-induced mechanical effects during a very short exposure time

SUMMARY:
Prospective, blinded, one arm, baseline-controlled clinical study for the evaluation of the UltraShape treatment for non-invasive abdominal fat reduction.

Study subjects will undergo UltraShape treatments on the abdominal area

DETAILED DESCRIPTION:
This study is a prospective, baseline and blinded controlled, one arm clinical study showing the performance and safety of the UltraShape treatment for non-invasive abdominal fat reduction.

Up to 60 Healthy subjects in up to 4 investigational sites will be enrolled in this study. All subjects will undergo an assessment of their general health. During the treatment period, subject's fat thickness and circumference will be measured and three successive UltraShape treatments, two weeks interval, will be performed.

The study subjects will undergo UltraShape treatments on the abdomen. During the follow-up period visit will be conducted as follow: 4 weeks (4wk FU), 8 weeks (8wk FU) and 12 weeks (12wk FU) post last treatment (Tx.3). Subject's abdominal fat thickness and circumference will be measured in the measurements points and will be assessed at each visit. Additionally, a subject questionnaire will be completed in each follow-up visit (4wk, 8wk and 12wk FU). Finally, photography will be performed under visible light conditions of the front, right, left and back view. Most of the assessments will occur at each of the visits (all treatments and all follow-up visits) to the clinic.

ELIGIBILITY:
Inclusion Criteria:

A subject is eligible to participate in the study if he/she meets all the following inclusion criteria:

1. Signed informed consent to participate in the study.
2. Female and male subjects, 18 and 60 years of age at the time of enrollment
3. Fitzpatrick Skin Type I to VI.
4. Fat thickness of at least 1.5 cm in the treated area (measured by calibrated caliper).
5. BMI interval: BMI between 22 to 30 (normal to overweight, but not obese).
6. If female, not pregnant or lactating, must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e. oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
7. In addition, negative urine pregnancy test as tested before each treatment and at the last follow-up visit for women with child-bearing potential (e.g. not menopause).
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
10. Willingness to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
11. Willing to have photographs and images taken of the treated areas to be used, de-identified in evaluations, publications and presentations

Exclusion Criteria:

A subject is not eligible for participation in this study if he or she meets any of the following exclusion criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker or defibrillator, abdominal aortic aneurism
2. Known hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions
4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone
6. Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction
7. Previous body contouring procedures in the treatment area within 12 months
8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
9. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
10. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
11. Very poor skin quality (i.e., severe laxity)
12. Abdominal wall diastasis or hernia on physical examination
13. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
14. Obesity (BMI above 30)
15. Childbirth within the last 12 months or breastfeeding women. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
16. Unstable weight within the last 6 months (i.e., ± 3 percent weight change in the prior six months)
17. Inability to comply with circumference measurement procedure (e.g., inability to hold breath for the required duration).
18. Fat thickness lower than 2.5 cm after strapping at the treated area.
19. Participation in another clinical study involving same anatomical areas within the last 6 months (or 30 days in case different anatomical areas were treated in previous trials).
20. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-06 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Abdominal fat thickness Reduction | 16 weeks
  Abdominal fat thickness Reduction post UltraShape treatments at 12 weeks follow-up (12wk FU) versus baseline

SECONDARY OUTCOMES:
Evaluate the safety of the treatment | day 0 until 16 weeks
  Evaluate the safety of the treatment with the UltraShape device on abdominal area
Abdominal fat thickness reduction as measured by Ultrasound | 8wk , 12wk , and 16wk
  Abdominal fat thickness reduction as measured by Ultrasound device post UltraShape treatments at all follow-up visits (4wk FU, 8wk FU, and 12wk FU) versus baseline
Abdominal fat thickness reduction as measured by caliper | 8wk , 12wk , and 16wk
  Abdominal fat thickness reduction as measured by caliper post UltraShape treatments at all follow-up visits (4wk FU, 8wk FU, and 12wk FU) versus baseline
Abdominal circumference reduction | 2 weeks , 4 weeks, 8wk , 12wk , and 16wk
  Abdominal circumference reduction post UltraShape treatments at all visits (treatments (pre Tx. 2; pre Tx.3) and follow up (4wk FU, 8wk FU, and 12wk FU)) versus baseline
Investigator satisfaction: | 8wk , 12wk , and 16wk
  Satisfaction assessment will be performed independently by the investigator himself using 5 points Likert scale questionnaire at all follow-up visits (4wk FU, 8wk FU and 12wk FU)
Subject satisfaction: | 8wk , 12wk , and 16wk
  Satisfaction assessment will be performed independently by the subject himself using 5 points Likert scale questionnaire at all follow-up visits (4wk FU, 8wk FU, and 12wk FU).
Comfort level during treatment: | day 0 , 2 weeks , 4 weeks
  Comfort assessment will be performed independently by the subject himself using a numerical scale. The subjects will answer this questionnaire after each of the three treatments

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Dover, M.D., Principal Investigator — SkinCare Physicians
Locations (2):
- United States (2):
  - Skin Care Physicians, Chestnut Hill, Massachusetts
  - Zel Skin & Laser Specialists, Edina, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hexsel D, Serra M, Mazzuco R, Dal'Forno T, Zechmeister D. Phosphatidylcholine in the treatment of localized fat. J Drugs Dermatol. 2003 Oct;2(5):511-8. PMID 14558399
- [Derived] Weinstein Velez M, Ibrahim O, Petrell K, Dover JS. Nonthermal Pulsed Ultrasound Treatment for the Reduction in Abdominal Fat: A Pilot Study. J Clin Aesthet Dermatol. 2018 Sep;11(9):32-36. Epub 2018 Sep 1. PMID 30319729